CLINICAL TRIAL: NCT06286722
Title: Optimized Rehabilitation of Older Adults With Hip Fracture and Signs of Cognitive Impairment - the ENHANCE Project - Feasibility Study
Brief Title: Optimized Rehabilitation of Older Adults With Hip Fracture and Signs of Cognitive Impairment - Feasibility Study
Acronym: ENHANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lolland Community, Denmark (Other)
Collaborators: Vordingborg Municipality (Unknown); Stevns Municipality (Unknown); Guldborgsund Municipality (Unknown); Frederiksberg Municipality (Unknown); Horsholm Municipality (Other)
Responsible Party: Principal Investigator, Mr. Jan Overgaard, Principal Investigator, Lolland Community, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LollandCD
Record Dates: First submitted 2024-02-07; First posted 2024-02-29 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hip Fractures; Cognitive Impairment
Keywords: Outpatient; Rehabilitation; Progressive; structured exercise; Hip Fracture; Cognitive impairment; Older adults
MeSH Terms: conditions — Hip Fractures; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Progressive, individualized and structured exercise program (Experimental): Individualized, progressive, structured exercise program. Participants will receive 12-weeks of either home-based and/or at a healthcare center intervention.
  The "at home" intervention will consist of 3 visits/sessions per week (approximately 30-60 min.) for 12 weeks (maximum of 36 sessions in total) delivered in the participants own home, temporary home (e.g. 24- hour rehabilitation facility), nursing home or assisted living facilities.
  The "at a healthcare center" intervention will be suggested to the participant when the physiotherapist and the participant feel confident that the participant can handle the transportation to/from the healthcare center, and will benefit from the higher intensity of the "at a healthcare center" intervention. This intervention consists of 2 visits/sessions per week (approximately 45-60 min.) for 12 weeks (total maximum of 24 sessions).
  Interventions: Other: Progressive, individualized and structured exercise program

INTERVENTIONS:
Other: Progressive, individualized and structured exercise program — See description under Arms

SUMMARY:
Older adults suffering from a hip fracture are a significant concern, with higher incidence rates among women. Mortality rates post-hip fracture are alarming, with up to 8-fold increased risk within 3 months and significant percentages within 30 days and 12 months. Older adults with hip fracture face challenges in regaining pre-fracture level of function, especially those with cognitive impairment, which affects 25% to 40% of cases and increases mortality risk. While interventions exist, such as progressive strength training and structured exercise programs, patients with hip fracture don't consistently restore pre-fracture function, particularly in cognitively impaired patients, who are often excluded from studies. Limited evidence exists on effective management for this subgroup, with a lack of clarity on community-based rehabilitation. Although guidelines suggest exercise interventions for patients with mild to moderate cognitive impairment, the specifics remain uncertain due to insufficient research focused solely on this population.

This feasibility study aims to assess the practicality and safety of implementing a 12-week individualized, progressive exercise program for older adults with hip fracture and cognitive impairment in an outpatient setting. Additionally, the investigators seek to gather qualitative insights through observations and interviews regarding participants' experiences and the perceived value of rehabilitation post-hip fracture, particularly focusing on the exercise intervention provided.

DETAILED DESCRIPTION:
Background and overall aim. Approximately 7,000 people suffer a hip fracture in Denmark each year. A hip fracture is a traumatic event with high mortality rates, and older adults with hip fractures experience significant pain, a general decline in functional ability, and difficulty regaining the same level of function (e.g., being able to move freely without walking aids) as before the fracture. Older adults with hip fracture and signs of cognitive impairment constitute a subgroup, accounting for 25-40% of the total group. Dementia increases the likelihood of sustaining a hip fracture nearly threefold and results in higher mortality rates compared to the rest of the patient group. Furthermore, many individuals do not receive the treatment/training they are entitled to, despite being initially worse off than those without signs of cognitive impairment. There is limited research in this area because older adults with signs of cognitive impairment are often excluded from research studies. The few studies available suggest that older adults with hip fracture and signs of cognitive impairment may benefit from the same interventions provided to older adults with hip fracture who do not have signs of cognitive impairment. However, no randomized controlled trials have been conducted to investigate whether a systematic, well-planned, and personalized home training program is superior to the standard training offered in municipalities for older adults with hip fracture and signs of cognitive impairment. With this feasibility study it is intended to assess the practicality and safety of a 12-week individualized, progressive exercise program for older adults with hip fracture and signs of cognitive impairment in a municipality-based setting shortly after discharge from hospital. Hopefully, and if there are positive results from this feasibility study the investigators will proceed with a randomized controlled trial (in another study).

ELIGIBILITY:
Inclusion Criteria:

* Recently (within 3 weeks) underwent surgical repair of a hip fracture (femoral neck or trochanteric fracture)
* Independent pre-fracture ambulatory function (≥2 on the New Mobility Score on indoor walking)
* Having signs of cognitive impairment measured with the Mini-Mental Score Examination of <24 points, or a verified dementia diagnosis, or on information from the patient record
* Living in their own home, nursing home, or assisted living facilities
* Informed consent by patient

Exclusion Criteria:

* Pathological hip fracture
* Having signs of severe dementia measured with the Mini-Mental State Examination (<10 points)
* Non-Danish speaking
* Patients with an unstable health condition (e.g. not treated high blood pressure (>180 mm HG)) evaluated by medical consultant
* "Safety concerns" (e.g. underlying comorbidities that might be associated with serious adverse events) - not safe to participate in the opinion of the investigator
* Having behavioral or psychotic disorders
* Alcohol or drug abuse
* Unable to participate in the intervention (e.g. due to blindness, no language)
* Patients with any weight-bearing restrictions after surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The New Mobility Score | Baseline, 3 months, 6 months
  The New Mobility Score is a composite score of the participant's ability to perform: indoor walking, outdoor walking and shopping, providing a score between zero and three (0: not at all, 1: with help from another person, 2: with an aid, 3: no difficulty) for each function, resulting in a total score from 0 to 9, with nine indicating a high functional level.

SECONDARY OUTCOMES:
Mini Mental State Examination | Baseline and 6 months
  A test to assess a participants cognitive level from a score from 0 to 30 points. A Mini-Mental State Examination can be used to check for cognitive impairment. The maximum score is 30 points. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.
Height | Baseline
  To assess the participants height in meters
Weight | Baseline, 3 months, 6 months
  To assess the participants weight in kilograms
Tandem balance test | Baseline, 3 months, 6 months
  A static balance test scoring the participants ability to stand in 3 different positions (0-30 point, where 30 points indicating no balance problem to 0 points = having seriously balance problems)
The Barthel-20 | Baseline, 3 months, 6 months
  To assess basic activities of daily living functions with the Barthel-20 test. Total possible scores range from 0-20, with lower scores indicating increased disability and higher score indicating independency.
30 sec chair raise test | Baseline, 3 months, 6 months
  This test examines the participants ability to raise up from a chair for as many times as possible within 30 seconds
Brief Assessment of Impaired Cognition Questionaire | Baseline, 3 months, 6 months
  A test to evaluate the participants cognitive level with a score ranging from 0 (= serious cognitive problems) to 20 point (= no impaired cognition).
Handgrip strength measurement | Baseline, 3 months, 6 months
  An assessment of the participants handgrip strength with a handheld grip strength dynamometer.
The Cumulated Ambulation Score | Baseline, 3 months, 6 months
  This score describes the participants independence in three activities (getting in and out of bed, sit-to-stand-to-sit from a chair, and walking). Each activity is assessed from 0-2 (0 = Not able to, despite human assistance and verbal cueing, 1 = Able to, with human assistance and/or verbal cueing from one or more persons, 2 = Able to safely, without human assistance or verbal cueing, use of a walking aid allowed). Total score ranging from zero to six points
Four meter walk test | Baseline, 3 months, 6 months
  To assess the participants gait speed over 4 meter walk.
Euroqol 5 dimensions | Baseline, 3 months, 6 months
  The Euroqol 5 dimensions essentially consists of 2 overall items; a descriptive system and the Euroqol visual analogue scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The Euroqol visual analog scale records the patient's self-rated health on a vertical visual analogue scale ranging from 0 to 100 with endpoints labelled 'The best health you can image' (= 100) and 'The worst health you can image' (= 0). The visual analog scale can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Clinical Frailty Scale | Baseline, 3 months, 6 months
  The Clinical Frailty Scale is a 9-point scale (ranging from 1 to 9) to summarize the overall level of fitness or frailty of an participant after they have been evaluated by a health care professional. The Clinical Frailty Scale is scored so that higher scores mean greater risk/frailty.
The Verbal Rating Scale | Baseline, 3 months, 6 months
  To assess the level of hip fracture-related pain using a 5 point scale (0 = no pain, 1 = light pain, 2 = moderate pain, 3 = severe pain, 4 = intolerable pain) in participants with hip fracture.
Activity accelerometers | Baseline, 3 months, 6 months
  To measure the amount of physical activity within 7 days. The two accelerometers (one placed on the wrist, the other on the thigh) will be monitor the participants activity level for 7 continous days (24 H a day).

CONTACTS AND LOCATIONS:
Overall Officials: Trine Nordentoft, Study Chair — Vordingborg Municipality; Halil Baldan, Study Chair — Guldborgsund Municipality; Lotte Bylov, Study Chair — Stevns Municipality; Gwen Tremmel, Study Chair — Lolland Municipality
Locations (6):
- Denmark (6):
  - Frederiksberg Healthcare center and 24-hour rehabilitation, Frederiksberg
  - Stevns Healthcare Center, Stevns Municipality, Hårlev
  - Hørsholm Health and Rehabilitation Center, Hørsholm
  - Maribo Health Center, Lolland Municipality, Maribo
  - Guldborgsund Healthcare Center, Guldborgsund Municipality, Nykøbing Falster
  - Vordingborg Healthcare Center, Vordingborg Municipality, Vordingborg